CLINICAL TRIAL: NCT02361814
Title: The Effect of Human Amniotic Membrane Allograft on Functional Recovery After Flexor Tendon Repair: a Pilot Study
Brief Title: The Effect of Human Amniotic Membrane Allograft on Functional Recovery After Flexor Tendon Repair
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unfavorable results
Sponsor: Tampere University (Other)
Collaborators: Tampere University Hospital (Other); Central Finland Hospital District (Other)
Responsible Party: Principal Investigator, Olli Leppänen, Researcher, Tampere University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R15002
Record Dates: First submitted 2015-02-03; First posted 2015-02-12 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Flexor Tendon Injury
Keywords: flexor tendon; finger; amniotic membrane; allograft; tendon injury
MeSH Terms: conditions — Tendon Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Amniotic membrane allograft group (Experimental): After the conventional flexor tendon repair, the amniotic membrane will be wrapped around the tendons and its borders will be fixed to the remaining tendon sheath.
  Interventions: Procedure: The use of amnionic membrane allograft

INTERVENTIONS:
Procedure: The use of amnionic membrane allograft — After the conventional flexor tendon repair, the amniotic membrane will be wrapped around the tendons and its borders will be fixed to the remaining tendon sheath.

SUMMARY:
The objective of this pilot study is to gain observational insight into potential preventive features of amniotic membrane transplantation in the adhesion formation after flexor tendon repair.

DETAILED DESCRIPTION:
The treatment of flexor tendon transection consists of surgical apposition of the lacerated tendon ends using non-absorbable sutures. Main complications which result in poor outcome of the tendon repair are the rupture of the tendon apposition or substantial adhesion formation between the two tendons or the tendon and the fibro-osseous canal. Adhesion formation is presumed to be a byproduct of the tendon healing. In the course of last 70 decades, the preventive effects of several pharmacological agents and mechanical barriers on adhesion formation have been investigated with some promising findings. One of the mechanical barriers that has been proposed to be suitable for adhesion prevention is human amniotic membrane allograft. However, there are no clinical studies evaluating the use of amniotic membrane in flexor tendon repair.

This is a pilot study for the forthcoming randomized controlled study. The objectives of the pilot study are: 1) to test the handleability of the human amniotic membrane allograft in flexor tendon sheath reconstruction in conjunction with flexor tendon repair, 2) to elucidate the possible adverse effects related to the use of amniotic membrane in flexor the sheath, and 3) to gain observational insight into potential preventive features of amniotic membrane transplantation in the adhesion formation. The hypothesis of the pilot study is that the application of the human amniotic membrane allograft in tendon sheath reconstruction in flexor tendon injury patients is technically feasible and results in no adverse effects to the patient.

A total of 10 patients with an acute flexor tendon injury will be included in the pilot study. After conventional tendoraphia, the amniotic membrane will be wrapped around the tendons and its borders will be fixed to the remaining tendon sheath. The primary outcome measure is total range of movement after 6 months of the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Acute flexor tendon transection in zone 2 in digits 2, 3, 4, or 5 (diagnosed within 1 week after the injury)
* Age over 18
* Patient's willingness to participate in the study

Exclusion Criteria:

* Tendon transection within 8 mm of its distal insertion (requiring reinsertion)
* Soft-tissue loss, severe crush, fracture, palmar plate injury, patient requiring revascularization
* Cognitive impairment or other factors (prisoner, military serviceman) which may affect one's decision making
* Substance abuse
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Total range of movement of the injured finger | 6 months

SECONDARY OUTCOMES:
Total range of movement of the injured finger | 2, 4, and 8 weeks
Rupture of the repair | 2, 4, 8 weeks, and 6 months
Postoperative infection | 2, 4, 8 weeks, and 6 months
QuickDASH -score | 2, 4, 8 weeks, and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Harry Göransson, M.D., Ph.D., Study Chair — Tampere University Hospital
Locations (1):
- University of Tampere, Tampere, Finland